CLINICAL TRIAL: NCT01499576
Title: Acetic Acid Chromoendoscopy for Judging Extent of Gastric Intestinal Metaplasia
Brief Title: Acetic Acid Chromoendoscopy to Judge Gastric Intestinal Metaplasia
Acronym: IM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konyang University Hospital (Other)
Responsible Party: Principal Investigator, Kyung Ho Song, MD, Assistant Professor, Konyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 11-62
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Stomach Neoplasms; Metaplasia
Keywords: Mass Screening; Endoscopy, Gastrointestinal; Stomach Neoplasms; Metaplasia; Diagnosis; Acetic acid; Chromoendoscopy
MeSH Terms: conditions — Stomach Neoplasms; Metaplasia; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acetic acid spraying (Experimental)
  Interventions: Procedure: Acetic acid chromoendoscopy

INTERVENTIONS:
Procedure: Acetic acid chromoendoscopy — Acetic acid chromoendoscopy Spraying 1.5% acetic acid(or vinegar), during screening gastroduodenoscopy

SUMMARY:
The presence and the extent of gastric intestinal metaplasia(IM) is a good indicator of high risk group of gastric cancer. Many methods was developed to survey it, including multiple gastric biopsy or methylene blue chromoendoscopy. But they are not practical in the routine screening exam, limited by cost and accessibility. Spraying of acetic acid is commonly used in screening cervical cancer, to induce whitish discoloration of metaplastic mucosa. The investigators have confirmed such whitish discoloration is induced in gastric IM, with accuracy > 80% in a pilot study of the investigators. This prospective study will tell the accuracy, sensitivity and specificity of acetic acid chromoendoscopy for judging gastric IM.

ELIGIBILITY:
Inclusion Criteria:

* Person who undergo gastroduodenoscopy
* Person who visit Konyang University Hospital

Exclusion Criteria:

* Bleeding diathesis
* History of stomach neoplasms
* History of upper gastrointestinal surgery

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Ho Song, M.D., Master, Principal Investigator — Konyang University
Locations (1):
- Department of Gastroenterology and Hepatology; Konyang University Hospital, Daejeon, South Korea

REFERENCES:
- [Background] Lambert R, Rey JF, Sankaranarayanan R. Magnification and chromoscopy with the acetic acid test. Endoscopy. 2003 May;35(5):437-45. doi: 10.1055/s-2003-38766. No abstract available. PMID 12701018
- [Background] Lee BE, Kim GH, Park DY, Kim DH, Jeon TY, Park SB, You HS, Ryu DY, Kim DU, Song GA. Acetic acid-indigo carmine chromoendoscopy for delineating early gastric cancers: its usefulness according to histological type. BMC Gastroenterol. 2010 Aug 23;10:97. doi: 10.1186/1471-230X-10-97. PMID 20731830
- [Background] Cassaro M, Rugge M, Gutierrez O, Leandro G, Graham DY, Genta RM. Topographic patterns of intestinal metaplasia and gastric cancer. Am J Gastroenterol. 2000 Jun;95(6):1431-8. doi: 10.1111/j.1572-0241.2000.02074.x. PMID 10894575
- [Derived] Song KH, Hwang JA, Kim SM, Ko HS, Kang MK, Ryu KH, Koo HS, Lee TH, Huh KC, Choi YW, Kang YW. Acetic acid chromoendoscopy for determining the extent of gastric intestinal metaplasia. Gastrointest Endosc. 2017 Feb;85(2):349-356. doi: 10.1016/j.gie.2016.07.064. Epub 2016 Aug 8. PMID 27515128
- See also: Konyang University Hospital, Web page — http://www.kyuh.co.kr

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: From Oct 2011 to Mar 2012. Recruiting institute: Konyang University Hospital, via the outpatient clinic or General Examination Center.
Groups:
- Acetic Acid Spraying: Underwent acetic acid chromoendoscopy, with spraying 1.5% acetic acid, during screening gastroduodenoscopy.
Period: Overall Study
Arm/Group | Acetic Acid Spraying
Started | 126
Completed | 105
Not Completed | 21
Not completed — Physician Decision | 12
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | Acetic Acid Spraying
Number analyzed (Participants) | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 96
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 53
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 105

OUTCOME MEASURES:

1. Primary Outcome: Percent Agreement Between Acetic Acid Chromoendoscopy and Endoscopic Biopsy
Description: Endoscopist judges the presence and the extent of gastric intestinal metaplasia during acetic acid chromoendoscopy. Endoscopist perform five endoscopic biopsies according to the protocol. The degree of agreement between the chromoendoscopy and the endoscopic biopsy is assessed as %.
Time Frame: 3 months after the completion of the study (a pathologist reviewed all the biopsy slide)
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Acetic Acid Spraying
Number analyzed (Participants) | 105
Number analyzed (lesions) | 525
percentage of lesions
  Overall Sensitivity | 78.5
  Overall Specificity | 94.4
  Overall Accuracy | 89.2
  Body Sensitivity | 67.1
  Body Specificity | 94.7
  Body Accuracy | 89.4
  Antrum Sensitivity | 80.9
  Antrum Specificity | 93.6
  Antrum Accuracy | 88.4
Statistical Analysis 1: Comparison: Acetic Acid Spraying; Test type: Superiority or Other; percent agreement = 89.2

2. Secondary Outcome: Agreement of Acetic Acid Chromoendoscopic Reading Between the Two Endoscopists
Description: The findings of chromoendoscopy will be interpretated by two endoscoipists (read as positive or negative finding) independently.
  We calculate the Kappa index of agreement for the acetic acid chromoendoscopy.
Time Frame: One month after the completion of the study
Measure: Number; unit: Kappa index of agreement
Units Other Than Participants: lesions
Groups:
- Acetic Acid Spraying: The same participants primary outcome analysed
Arm/Group | Acetic Acid Spraying
Number analyzed (Participants) | 105
Number analyzed (lesions) | 505
Kappa index of agreement | 0.808
Statistical Analysis 1: Comparison: Acetic Acid Spraying; Test type: Superiority or Other; p < 0.01, Kappa index of agreement; Kappa index of agreement = 0.808

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events. Assess kind of side effect and severity. Measured by interview with a physician, just after the procedure and 1weak later.
Time Frame: up to 1week after the acetic acid chromoendoscopy
Measure: Number; unit: participants
Arm/Group | Acetic Acid Spraying
Number analyzed (Participants) | 105
participants
  Epigastric discomfort | 9
  Neck discomfort | 2
Statistical Analysis 1: Comparison: Acetic Acid Spraying; Test type: Superiority or Other; persent of adverse event = 10.48

ADVERSE EVENTS:
Arm/Group | Acetic Acid Spraying
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 11/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acetic Acid Spraying (N=105)
Epigastric discomfort (Gastrointestinal disorders) | 9
Odynophagia (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
Concomitant comparison with methylene blue chromoendoscopy was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No